CLINICAL TRIAL: NCT05616806
Title: Project LIGHT - Long COVID-19 Intervention Using Digital Health & Technology
Brief Title: Long COVID-19 Intervention Using Digital Health & Technology
Acronym: LIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022003396
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-11

CONDITIONS: Long COVID; Distress Tolerance
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- distress tolerance skills training (Experimental): technology delivered distress tolerance skills training
  Interventions: Behavioral: iENDURE

INTERVENTIONS:
Behavioral: iENDURE — Two delivery modes: computer and text message. The intervention provides introductory strategies for managing physical and emotional distress associated with Long COVID through a computer-delivered session followed by 4-weeks of theoretically-informed text messages intended to promote distress tolerance (DT).
  Computer - the initial intervention will be delivered online via the Qualtrics survey tool following informed consent. The intervention provides strategies to better tolerate emotional and physical discomfort to persist with behavioral goals. Text Message - The text message intervention will be delivered using Marigold Health (a HIPAA compliant platform for secure text messaging). Participants will receive daily text messages that focus on emphasizing adaptive strategies for tolerating physical and emotional discomfort in order to work toward behavioral goals. The text messages will be personalized and offer skills training (reminders of previously learned DT skills).
  Other Names: Marigold Health

SUMMARY:
The current study seeks to pilot test the iENDURE (Enhancing Distress tolerance to Uplift motivation in Recovery) intervention among 10 participants with Long COVID (Coronavirus Disease) symptoms. Following informed consent procedures, participants will complete a brief baseline assessment of self-report measures. Participants will then engage in the iENDURE intervention (described below) for 4 weeks. At the end of the intervention period, participants will complete another brief assessment of self-report measures and a qualitative interview about their experience with the program. Participants will be compensated for completing the baseline and post-intervention assessments

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age
* Must speak English proficiently
* Must own a text-enabled device
* Diagnosis (self-reported) of COVID-19
* Diagnosis (self-reported) of Long-COVID symptom(s)
* Must be able to provide written, informed consent

Exclusion Criteria:

* Not fluent in English
* Limited mental capacity or inability to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Score (CSQ-8) | 4 weeks
  Measure satisfaction scores after 4 weeks of using the intervention for this group of participants with Long COVID as measured by the client satisfaction questionnaire. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
System Usability Score (SUS) | 4 weeks
  Measure usability after 4 weeks for this group of participants with Long COVID as measured by the 10 item system usability scale. In the SUS instrument, even and odd questions are scored differently. Odd questions are scored 0-4 based on the 1-5 selection, where a selection of 1 equals 0 points, a selection of 2 equals 1 point, and so on. Even questions are scored 4-0 on the 1-5 selection where a selection of 1 equals 4 points, a selection of 2 equals 3 points, and so on. Scores for all ten questions are added up for a total score between 0-40 points. This total is multiplied by 2.5 to generate a SUS score between 0-100 points. Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Langdon, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No